CLINICAL TRIAL: NCT04794985
Title: Post-COVID-Health Study: Multidimensional Health Status of COVID-19 Survivors One Year After a SARS-CoV-2 Infection
Status: Terminated | Type: Observational
Why Stopped: With included subjects (n=140) we have sufficient power to answer the primary research question.
Sponsor: Maastricht University Medical Center (Other)
Collaborators: VieCuri Medical Centre (Other); Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: NL76949.068.21
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Covid19
Keywords: Multidimensional health; COVID-19; Long-term consequences
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood samples will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study assesses the multidimensional health status of COVID-19 survivors one-year post-infection using validated subjective and objective measures.

DETAILED DESCRIPTION:
Rationale: Within the Netherlands, more than 1 million people have been infected with SARS-CoV-2, also known as COVID-19. Although the mortality rate is considerable, the vast majority of COVID-19 patients survive the infection. Preliminary findings show that a majority of COVID-19 survivors still experience health problems 3 months after the infection, including reduced lung diffusion capacity, low exercise capacity, muscle weakness, mental problems and reduced cognitive function resulting in a generally poor health status. Whether these health consequences persist on the long-term is unknown.

Objective: To assess the multidimensional health status of COVID-19 survivors one-year post-infection using validated subjective and objective measures.

Study design: A multicenter prospective observational study performed within the MUMC+ and VieCuri Medical Center.

Study population: 200 COVID-19 survivors of the MUMC+, VieCuri Medical Center or Zuyderland Medical Center, both hospitalized (ICU and non-ICU admitted) as well as non-hospitalized patients.

Main study parameters/endpoints: Outcome parameters include objectively and subjectively measured multidimensional health outcomes including physiological and metabolic health, physical capability, cognitive function, psychosocial well-being, social well-being, patient reported outcomes as well as potential determinants of these multidimensional health outcomes (e.g. treatment during/after SARS-CoV-2 infection, vaccination, comorbidities, medication use etc.). Outcomes will be measured during a one-day study visit.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects will benefit from participating within this study, because their general health will be evaluated in detail and from a multidimensional perspective. Furthermore, subjects will be informed on their multidimensional health outcomes and will receive a lifestyle advice tailored to their health status. Risks and inconveniences are limited to the time investment associated with the completion of the questionnaires and the study visit. During the study visit various non-invasive measurements as well as minor invasive blood sampling will be performed.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive based on:

  * Confirmed RT-PCR;
  * Proven serology for SARS-COV-2 with clearly associated complaints for a SARS-COV-2 infection;
  * CO-RADS score of 4 or more with a proven serology for SARS-CoV-2 afterwards.
* Age of ≥18 years;
* Able to provide informed consent;
* Understanding of Dutch language.

Exclusion Criteria:

* Patients not willing to participate;
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All COVID-19 survivors of the MUMC+, VieCuri Medical Center or Zuyderland Medical Center can be included in this study. Both hospitalized (ICU and non-ICU admitted) as well as non-hospitalized patients will be eligible for participation.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Lung function measured with spirometry | 1 year post-infection
  Pre- and post-bronchodilator spirometry will be performed to determine forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1).
Diffusion capacity measured with the single breath method | 1 year post-infection
  To determine diffusion capacity for carbon monoxide
(Persistent) lung damage | 1 year post-infection
  To determine lung damage a chest CT-scan will be obtained. To evaluate whether lung damage is persistent, scans will be compared to scans obtained during COVID-19 screening or COVID-19 after care.
Bone mineral density by dual-energy X-ray (DEXA)-scan | 1 year post-infection
  Total bone mineral density (BMD) as well as BMD of the lumbar spine and total hip-neck will be determined using a DEXA-scan.
Lean mass by dual-energy X-ray (DEXA)-scan | 1 year post-infection
  Total lean mass will be determined using a DEXA-scan.
Fat free mass by dual-energy X-ray (DEXA)-scan | 1 year post-infection
  Total fat free mass will be measured using a DEXA-scan.
Fat mass by dual-energy X-ray (DEXA)-scan | 1 year post-infection
  Total fat mass and fat percentage as well as visceral fat mass will be measured using a DEXA-scan.
Vertebral fracture assessment by dual-energy X-ray (DEXA-scan) | 1 year post-infection
  Vertebral fracture assessment will be determined using a DEXA-scan.
Muscle cross sectional area on chest CT-scan | 1 year post-infection
  Muscle cross sectional area will be determined based on pre-established Hounsfield Units on the chest CT-scan.
Adipose tissue cross sectional area on chest CT-scan | 1 year post-infection
  Muscle cross sectional area will be determined based on pre-established Hounsfield Units on the chest CT-scan.
Weight will be measured on a weighing scale | 1 year post-infection
  Weight will be measured on a weighing scale.
Height will be measured using a stadiometer | 1 year post-infection
  Height will be measured using a stadiometer.
Body mass index (BMI) will be calculated from the weight and height | 1 year post-infection
  Weight and height will be combined to report BMI in (kg/m^2)
Fasted resting energy expenditure by indirect calorimetry (ventilated hood) | 1 year post-infection
  VO2 and VCO2 will be measured to determine energy expenditure.
Resting blood pressure | 1 year post-infection
  Resting diastolic and systolic blood pressure will be measured as part of the cardiometabolic profile to determine the prevalence of the metabolic syndrome.
Waist circumference | 1 year post-infection
  Waist circumference will be measured as part of the cardiometabolic profile to determine the prevalence of the metabolic syndrome.
Fasting glucose levels | 1 year post-infection
  Fasting glucose levels will be determined in sampled blood as part of the cardiometabolic profile to determine the prevalence of the metabolic syndrome.
Fasted lipid profile | 1 year post-infection
  Fasted high-density, low-density and total lipoprotein levels (HDL and LDL) as well as triglycerides will be measured as part of the cardiometabolic profile to determine the prevalence of the metabolic syndrome.
Six minute walking test to determine exercise capacity | 1 year post-infection
  Six minute walking distance will be determined.
Peak work rate by cardiopulmonary cycling exercise test (CPET) | 1 year post-infection
  Maximal work rate (W) will be determined during the CPET
Peak O2-consumption and CO2-production by cardiopulmonary cycling exercise test (CPET) | 1 year post-infection
  Maximal O2 consumption and CO2 production will be determined during the CPET.
Maximal heart rate during cardiopulmonary cycling exercise test (CPET) | 1 year post-infection
  Maximal heart will be measured during the CPET.
Respiratory muscle strength by mouth pressure | 1 year post-infection
  Inspiratory and expiratory mouth pressure will be measured.
Upper extremity muscle strength by measuring handgrip strength | 1 year post-infection
  A hydraulic grip strength dynamometer will be used to measure the maximal handgrip strength.
Lower extremity muscle strength by measuring isometric muscle strength | 1 year post-infection
  Maximal isometric upper leg muscle strength will be measured of the quadriceps muscle using a Biodex dynamometer.
Mobility using the short physical performance battery (SPPB) | 1 year post-infection
  The SPPB consists of three types of physical maneuvers: the balance test, the gait speed test and the chair stand test leading to a score of 0-12. Lower scores indicate less mobility.
Physical activity level by accelerometry | 1 year post-infection
  An accelerometer will be worn for 7 days to determine physical activity level.
Cognitive function by Montreal Cognitive Assessment (MOCA) | 1 year post-infection
  The MOCA will lead to a total score of 0-30, in which lower scores indicate less cognitive function.
Cognitive function using the cognitive failure questionnaire (CFQ) | 1 year post-infection
  The CFQ will lead to a total score of 0-100. A higher total score indicates more subjective cognitive failure. Additionally, four subscales can be identified, related to distraction, distraction in social situations, names and words and orientation.
Dietary intake by a food diary | 1 year post-infection
  A 3-day food diary will be used to investigate the dietary intake.
Smell by the Sniffing Sticks treshold test | 1 year post-infection
  The average of the last four reversal points is used as final threshold score.
Taste using the taste strips 'filter paper disc method' test | 1 year post-infection
  A maximum score of 16 correct taste detections can be retrieved indication good taste function.
Taste and smell function using the taste and smell function questionnaire | 1 year post-infection
  The questionnaire will retrieve a maximal score of 0-52 and 0-44 for taste and smell, respectively, in which higher scores indicate problems with taste and smell function.
The hospital anxiety and depression scale (HADS) to determine anxiety and depression levels | 1 year post-infection
  The HADS will retrieve a total score of 0-21 in which lower levels indicate higher levels of anxiety or depression.
The Perceived stress scale (PSS) to determine stress levels | 1 year post-infection
  The PSS will retrieve a total score of 0-40 in which lower scores indicate higher stress levels.
Perceived social support using the multidimensional scale of perceived social support (MSPSS) | 1 year post-infection
  A total score of 12-84 can be retrieved in which lower scores indicate lower levels of social support.
Loneliness using the loneliness scale (LS) | 1 year post-infection
  The LS will retrieve a total score of 0-11 in which higher scores indicate strong loneliness.
Subjective multidimensional health status by euroqol-5 dimensions | 1 year post-infection
  The EQ-5D consists of 5 domains (mobility, self-care, usual activity, pain/discomfort, anxiety/depression) and a visual analogue scale.
Dyspnea using the modified medical research council (mMRC) | 1 year post-infection
  The mMRC will retrieve a total score of 0-5 in which higher levels indicate more dyspnea.
Fatigue using the Checklist Individual Strength (CIS) | 1 year post-infection
  The CIS will retrieve a total score of 20-140 in which higher scores indicate more fatigue.
Sleep quality using the Pittsburgh Sleep Quality Index (PSQI) | 1 year post-infection
  The total PSQI score will vary between 0-21 in which higher scores indicate poor sleep quality.
General pain using the Visual Analogue Scale (VAS) | 1 year post-infection
  A total score of 0-100 will be retrieved in which higher scores indicate more pain.

SECONDARY OUTCOMES:
Medical history | 1 year post-infection
  Retrieved from medical records and self-report
Treatments/therapies after SARS-CoV-2 infection | 1 year post-infection
  Retrieved from medical records and self-report
Vaccination for COVID-19 | 1 year post-infection
  Retrieved from medical records and self-report
Re-infection with COVID-19 | 1 year post-infection
  Retrieved from medical records and self-report
Medication use | 1 year post-infection
  Retrieved from medical records and self-report

OTHER OUTCOMES:
Smoking status | 1 year post-infection
  Based on self-report
Sociodemographics | 1 year post-infection
  Including age, gender, race, living situation, household composition, marital status, educational level, smoking status, alcohol consumed, employment status, occupation, volunteer work, and income level.
Motivation by the Behavioral Regulation in Exercise Questionnaire (BREQ-2) | 1 year post-infection
  The BREQ-2 will provide several motivation types based on the self-determination theory.
Motivation by the Regulation of Eating Behaviors Questionnaire (REBS) | 1 year post-infection
  The REBS will provide several motivation types based on the self-determination theory.
Date of SARS-CoV-2 infection | 1 year post-infection
  The date of the SARS-CoV-2 infection will be extracted from the medical records in order to determine the time since the COVID-19 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Schols, PhD, Study Director — Maastricht University Medical Centre
Locations (3):
- Netherlands (3):
  - Zuyderland Medical Center, Heerlen
  - Maastricht University Medical Center, Maastricht
  - VieCuri Medical Center, Venlo

IPD SHARING:
Plan to Share IPD: Undecided